CLINICAL TRIAL: NCT05026580
Title: Long-term Changes in Health Outcomes During Digitally Delivered Exercise and Education Treatment for Hip and Knee Osteoarthritis
Brief Title: Outcomes During Digitally Delivered Osteoarthritis Treatment
Status: Withdrawn | Type: Observational
Why Stopped: Study halted due to unforeseen challenges in securing the necessary resources to conduct the research effectively.
Sponsor: Joint Academy (Industry)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: EQ-5D-5L
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Health-related Quality of Life; Pain; Function; Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Osteoarthritis; Exercise; Digital; Telehealth; Physiotherapy
MeSH Terms: conditions — Pain; Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Joint Academy exercise and education smart phone application — The Joint Academy® (www.jointacademy.com) program for people with hip or knee OA consists of video instructed and progressively adaptable daily exercises, patient education through text lessons and a continuous asynchronous chat function with a personal reg. physiotherapist who supervises the patient during the full participation period.

SUMMARY:
Objectives: To examine changes in health-related quality of life (HRQL), pain and function among patients with knee or hip osteoarthritis (OA) participating in digitally delivered exercise and education treatment for up to 12 or 24 month.

Design: An observational longitudinal and repeated cross-sectional cohort study.

Investigators will include participants who have participated in the digitally delivered exercise and education treatment program Joint Academy® for 3, 6 , 9 , 12 and if enough patients also for 24 month. Investigators will analyze both cross-sectional samples at each time point and a longitudinal sample that have participated for at least 12 month, with at least one follow-up in between.

Outcomes: Investigators will analyze HRQL with EQ-5D-5L, pain with Numeric Rating Scale (NRS) 0-10 (best to worst) and function with 30-sec chair stand test (CST) at baseline and at 3, 6, 9,12 and if possible 24 months during the treatment. Main outcome will be change in level in EQ-5D-5L dimensions. We will also analyze minimally clinical important changes (improved or not) and mean changes in EQ-5D-5L index score, pain and 30-sec chair stand test (CST). Logistic regression models and linear mixed models will be used for analysis. Analyses will be performed for repeated cross-sectional samples and a longitudinal sample.

DETAILED DESCRIPTION:
International treatment guidelines recommend exercise, education and weight control (if needed) as first-line treatment for knee and hip osteoarthritis (OA). Still, evidence suggest that less than 50% of OA patients have participated in first-line treatment before getting joint replacement.

Several observational and randomised controlled trials (RCTs) show that exercise therapy is effective in reducing pain, improving physical function and health-related quality of life (HRQL) at clinically important levels in the short-term.

Quality of life is rated lower by people with OA compared to norm populations and measures of well-being are increasingly used as outcomes in health interventions. Face-to-face first-line OA treatment following the Better Care for persons with OsteoArthritis (BOA) or Good Life with osteoArthritis in Denmark (GLA:D) initiatives seem to have small but clinically significant effects on HRQL immediate after intervention, at six month and with maintained improvements at one year for knee but not hip OA.

The digitally delivered first-line OA treatment program Joint Academy® (JA) was developed in Sweden in 2016 in an attempt to improve implementation and adherence to guidelines. The program is based on evidence from BOA. Initial observational studies show that both patients with hip and knee OA had clinically important improvements in pain and function at six weeks with sustained improvements up to 48 weeks of treatment. Further, HRQL dimensions mobility and pain/discomfort significantly improved after six weeks, while others did not (self-care, usual activities, and anxiety/depression. However, the long-term change in HRQL during digitally delivered first-line OA treatment is not known.

Therefore, the aim is to identify changes in HRQL, pain and function, during up to12 months of digitally delivered first-line treatment. A second aim was to examine if changes differs between hip/knee and women/men.

Outcomes Outcomes were collected at start and at standardized time points during the treatment. They were chosen based on the International Consortium for Health Outcomes Measurement Standard Set for Hip & Knee Osteoarthritis (ICHOM), self-entered using the digital program interface and stored in the JA database.

HRQL was evaluated every third month using the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L), which is a generic quality of life measurement tool. The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. The levels of severity range from no problems (1) to extreme problems/unable to (5) and are recorded for each of the five dimensions. The raw scores are also converted to a single EQ-5D index value using a scoring algorithm (British tariff was used) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state). A change of ≥0.03 in the index was considered as minimally clinical important change (MCIC) according to a comprehensive review of musculoskeletal disorders.

Joint pain was assessed using the Numerical Rating Scale (NRS), with the instruction Mark on this scale how much pain you had the last week in your hip/knee, followed by a 0-10 scale where 0 indicates No pain and 10 indicates Maximum pain. A difference of 15 of 100 for absolute improvement (slightly or moderately) is considered as MCIC.

Physical function was assessed with the 30-s chair-stand test (CST) performed by the participant with the help of an instruction video with a coupled visual timer. The patient entered the performed number of repetitions after each test. The 30-s CST is recommended by the Osteoarthritis Research Society International (OARSI) as a performance-based functional test for knee and hip OA (Dobson 2013). A difference of two rises is considered as MCIC.

Data on the participants' overall health and characteristics such as OA location (hip/knee), age, sex, educational level (), height, weight and medical conditions (xx) were collected at inclusion.

ELIGIBILITY:
* Patients that had participated in the Joint Academy treatment program and given their informed consent
* Radiographic and or clinical diagnosis of hip or knee OA from a physical therapist or physician (95% of all patients in previously published studies). Individuals without a prior diagnosis had clinical OA confirmed by an orthopaedic surgeon or physiotherapist via telephone (diagnosis according to NICE criteria and Swedish National Guidelines, and confirming the absence of any red flag symptoms), or if deemed necessary were recommended to seek face-to-face care before inclusion in the programme.
* From October 1st 2021, all patients should have undergone a physical examination by doctor or physiotherapists before being able to enter the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants join the digital OA treatment program via online advertisements and campaigns placed on search engines and social networks, or by recommendations by their local physiotherapist or orthopaedic surgeon. Procedure for inclusion and exclusion has been described above. Data will be extracted from the Joint Academy (JA) database registry for Swedish patients who had started their treatment Janurary 1st 2019 or after. A
  Outcome analysis will be made for three different age groups.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | one year
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. The levels of severity for each dimension ranges from no problems (1) to extreme problems/unable to perform. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)

SECONDARY OUTCOMES:
Pain assessed with a Numeric Rating Scale (NRS) | one year
  Mark on this scale how much pain you had the last week in your hip/knee, followed by a 0-10 scale where 0 indicates No pain and 10 indicates Maximum pain
Physical function with the 30-sec chair stand test (CST) | one year
  The test is is the maximum number of repetitions of chair rises the participant can perform in 30 secords. It is performed by the participant with the help of an instruction video with a coupled visual timer

CONTACTS AND LOCATIONS:
Locations (1):
- Joint Academy, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided